CLINICAL TRIAL: NCT06598345
Title: Impact of Integrated Pet Care on Glycemic Control and Diabetes Responsibility
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00115936
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes Mellitis
Keywords: type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pet Fish with Integrated Diabetes Care + Collaborative Communication (Experimental): Participants will receive specific instructions for coupling daily and weekly fish care and diabetes care throughout the 12-week intervention and how to conduct weekly collaborative communication meetings.
  Interventions: Behavioral: Routine Pet Fish Care; Behavioral: Collaborative Communication
- Pet Fish with Integrated Diabetes Care Only (Active Comparator): Participants in the Pet Fish with Integrated Diabetes Care Only Group will be provided specific instructions for coupling the fish care and diabetes care throughout the 12-week intervention.
  Interventions: Behavioral: Routine Pet Fish Care
- Control (No Intervention): Participants in the Control Group will be told to monitor BG (blood glucose) four times daily, review BG readings with their parent weekly and document on their device's software.

INTERVENTIONS:
Behavioral: Routine Pet Fish Care — Participants in the Routine Group will be provided specific instructions for coupling the daily and weekly fish care and diabetes care throughout the 12-week intervention They will also be told to monitor BG four times daily, review BG readings with their parent weekly and document the BG checks and weekly reviews on their device's software.
  Arms: Pet Fish with Integrated Diabetes Care + Collaborative Communication; Pet Fish with Integrated Diabetes Care Only
Behavioral: Collaborative Communication — Parents and participants in the Collaborative Communication group will be given recommendations for how to conduct weekly meetings in a collaborative approach based on a modified version of the Minute Meeting protocol.
  Arms: Pet Fish with Integrated Diabetes Care + Collaborative Communication

SUMMARY:
The goal of this clinical trial is to learn if incorporating the structured care of a pet fish into a family-based diabetes self-care routine combined with communication skills training works to improve glycemic control, blood glucose monitoring frequency and blood glucose review in early adolescents with suboptimal control of type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* age 10-13 years (inclusive)
* diagnosis of T1DM for at least one year
* fluency in English or Spanish, (d) recent HbA1c value 7.5% - 14%
* utilization of a CGM or glucometer that links with software to enable viewing and documentation in daily report including a section to enter "notes" (i.e. CGM/software, Dexcom/Clarity; Freestyle Libre/LibreView; AccuChek,OneTouch (glucometers)/MySugr)
* current pet fish at home or willingness to obtain a pet fish if randomized to that intervention.

Exclusion Criteria:

* clinical or laboratory characteristics suggestive of type 2 DM
* involvement in foster care
* dual-home living situation
* severe psychiatric disorders
* developmental delay or cognitive impairment that make it difficult to establish consistent diabetes and pet care behaviors
* current participation in another study that may impact glycemic control
* HbA1c >14% (because these individuals may need a more intensive intervention than this is intended to provide)
* lack of a computer or compatible cell phone for uploading CGM or glucometer data.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Baseline
  Recruitment rate will be calculated as [number of participants assenting] divided by [number who were invited]
Fidelity to BGM (blood glucose monitoring) partnered with fish feeding | 3 months
  Fidelity to BGM partnered with fish feeding will be assessed by calculating the percentage of BG checks that were partnered with fish feeding.
Fidelity to weekly reviews partnered with fish tank maintenance | 3 months
  Fidelity to weekly reviews partnered with fish tank maintenance will be assessed by calculating the percentage of BG (blood glucose) reviews that were partnered with tank maintenance. The research team will review the data uploads on a weekly basis.
Retention rate | 3 months
  Retention rate will be calculated as [number of participants who continue fish care tasks] divided by [number who were eligible upon completion of the baseline assessment].

SECONDARY OUTCOMES:
Number of blood glucose (BG) readings receiving parental review | Baseline, during intervention and post-intervention (monthly intervals, up to 6 months)
  Weekly BG review will be determined using the Weekly Review notations on the device's digital platform.
Time in Range (TIR) | Baseline, 3 months, 6 months
  Time in range (TIR) for participants using a continuous glucose monitor will be expressed as percentage of glucose readings between 70-180 mg/dL for the 2 weeks prior to the study visit per the report (i.e. Dexcom Clarity®) which is downloaded in clinic as standard of care.
Self Care Inventory (SCI) (modified) | Baseline, 3 months, 6 months
  Three items from this validated measure assessing perceptions of adherence to diabetes self-care recommendations (BGM, BG review, insulin adjustment) over the previous 4 weeks will be used. Responses are on a 5-point Likert scale ranging from 0 = "Never do it" to 4 = "Always do this as recommended without fail".
Blood glucose monitoring (BGM) frequency | Baseline, 3 months, 6 months
  Daily BGM frequency will be determined using the BG notations on device's digital platform. The percentage of days on which participants complete four SMBGs (self-monitoring of blood glucose) will be reported.
HbA1c (Hemoglobin A1C) level | Baseline, 3 months, 6 months
  HbA1c is a biomarker that provides an estimate of glycemic control over the previous 3 months. HbA1c will be measured using a finger stick blood sample analyzed on a DCA Vantage Analyzer (Siemens). ADA recommends a goal of HbA1c <7% for this early adolescent age group.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Gupta, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No